CLINICAL TRIAL: NCT02277028
Title: A Comparison of Two Types of Priming for Upper Extremity Hemiparesis
Brief Title: Bilateral Priming for Upper Extremity Hemiparesis in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AOTFIRG13STOYKOV
Record Dates: First submitted 2014-10-24; First posted 2014-10-28 (Estimated); Results first posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-01

CONDITIONS: Stroke, Upper Extremity Hemiparesis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bilateral Priming (Experimental): Bilateral priming a priming technique which is non-invasive and free of side effects. The technique described in this study uses bilateral, symmetrical, rhythmic movement "bilateral priming" and its purpose is to ready the motor cortex for functional limb training. A "rocker" is used so that the less affected limb can drive the affected one in symmetrical wrist flexion and extension.
  There are 2 parts to this behavioral intervention. Bilateral priming and task specific training Dosage: 15 minutes of bilateral priming per day 3/days per week for 5/wks. Also 45 minutes of task specific training is delivered 3/days per week for 5/wks. The total of 30 hours of a combination of bilateral priming and task specific training can be completed within 6 weeks.
  Dosage frequency 2 times per day. Dosage type: Research participant must perform activities with hands as directed by an occupational therapist
  Interventions: Behavioral: priming and task specific training
- Health Education (Active Comparator): The group with no priming will receive stroke related health education via a website from the American Heart Association (15 minutes). They will use their affected hand (as they are able) This will be followed by 45 minutes of the same task specific arm training protocol described in the bilateral priming group. This group will follow the same schedule as experimental.
  There are 2 parts to this behavioral intervention. Computerized health education training and task specific training Dosage: 15 minutes of health education per day 3/days per week for 5/wks. Also 45 minutes of task specific training is delivered 3/days per week for 5/wks. A total of 30 hours of a combination of computerized stroke health education and task specific training can be completed within 6 weeks.
  Dosage frequency 2 times per day. Dosage type: Research participant must perform computerized health education activities with hands as well as task specific training directed by an occupational therapist
  Interventions: Behavioral: priming and task specific training

INTERVENTIONS:
Behavioral: priming and task specific training — This task specific training protocol has been used in several clinical trials.

SUMMARY:
This study will compare bilateral priming followed by task specific training to health care education followed by the same task specific training protocol. The intention is to understand the effects of priming on upper limb training post-stroke.

DETAILED DESCRIPTION:
Techniques to enhance use dependent plasticity have been examined in stroke rehabilitation research. The purpose of these techniques is to prime the cortex prior to training. The priming techniques previously described in the literature include medication (i.e. amphetamines), transcranial electric or magnetic stimulation, and manipulation of somatosensory input. Here, the investigators examine a priming technique which is non-invasive and free of side effects. The technique described in this study uses bilateral, symmetrical, rhythmic movement "bilateral priming" and its purpose is to ready the motor cortex for functional limb training. A "rocker" is used so that the less affected limb can drive the affected one in symmetrical wrist flexion and extension. In this project, the investigators intend to compare bilateral upper limb priming with task specfiic training to a health care education website program followed by the same task specific training as the experimental group.This active comparator (health care education) will receive stroke related health education via a website from the American Heart Association. Transcranial Magnetic Stimulation willl include measurement of transcallosal inhibition persistence from the affected hemisphere to the less affected hemisphere and vice versa ( less affected to affected). The investigators expect the bilateral priming group to have greater changes in transcranial magnetic stimulation measures and greater improvements in behavioral measures at all time points.

ELIGIBILITY:
Inclusion Criteria:

* Must have survived a unilateral stroke at least six months prior to enrollment
* Fugl Meyer Upper Extremity Score between 22-38.

Exclusion Criteria:

* No individuals who have a pacemaker, metal implant in head or neck, history of seizures, recent concussion or history of headaches

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Stoykov, PhD, Principal Investigator — Rush University
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] King EC, Doherty M, Corcos D, Stoykov ME. Examining recruitment feasibility and related outcomes in adults post-stroke. Pilot Feasibility Stud. 2020 Oct 24;6:160. doi: 10.1186/s40814-020-00696-w. eCollection 2020. PMID 33110623
- [Derived] Stoykov ME, King E, David FJ, Vatinno A, Fogg L, Corcos DM. Bilateral motor priming for post stroke upper extremity hemiparesis: A randomized pilot study. Restor Neurol Neurosci. 2020;38(1):11-22. doi: 10.3233/RNN-190943. PMID 31609714

RESULTS

PARTICIPANT FLOW:
Groups:
- Health Education: The group with no priming will receive stroke related health education via a website from the American Heart Association (15 minutes). They will use their affected hand (as they are able) This will be followed by 45 minutes of the same task specific arm training protocol described in the bilateral priming group. This group will follow the same schedule as above. The health education (15 minutes) will be following by task specific training (45 minutes). Subjects will then have a break (betw. 30-60 minutes) and then repeat the above. Total time on health education website for one day is 30 minutes. Total task specific training for one day is 90 minutes
  priming and task specific training: This task specific training protocol has been used in several clinical trials.
  8
- Bilateral Priming: Bilateral priming a priming technique which is non-invasive and free of side effects. The technique described in this study uses bilateral, symmetrical, rhythmic movement "bilateral priming" and its purpose is to ready the motor cortex for functional limb training. A "rocker" is used so that the less affected limb can drive the affected one in symmetrical wrist flexion and extension. The priming (15 minutes) will be following by task specific training (45 minutes). Subjects will then have a break (betw. 30-60 minutes) and then repeat the above. Total priming for one day is 30 minutes. Total task specific training for one day is 90 minutes
  priming and task specific training: This task specific training protocol has been used in several clinical trials.
  8
Period: Overall Study
Arm/Group | Health Education | Bilateral Priming
Started | 8 | 8
Completed | 7 | 7
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Bilateral Priming: Bilateral priming a priming technique which is non-invasive and free of side effects. The technique described in this study uses bilateral, symmetrical, rhythmic movement "bilateral priming" and its purpose is to ready the motor cortex for functional limb training. A "rocker" is used so that the less affected limb can drive the affected one in symmetrical wrist flexion and extension. The priming (15 minutes) will be following by task specific training (45 minutes). Subjects will then have a break (betw. 30-60 minutes) and then repeat the above. Total priming for one day is 30 minutes. Total task specific training for one day is 90 minutes
  priming and task specific training: This task specific training protocol has been used in several clinical trials.
- Health Education: The group with no priming will receive stroke related health education via a website from the American Heart Association (15 minutes). They will use their affected hand (as they are able) This will be followed by 45 minutes of the same task specific arm training protocol described in the bilateral priming group. This group will follow the same schedule as above. The health education (15 minutes) will be following by task specific training (45 minutes). Subjects will then have a break (betw. 30-60 minutes) and then repeat the above. Total time on health education website for one day is 30 minutes. Total task specific training for one day is 90 minutes
  priming and task specific training: This task specific training protocol has been used in several clinical trials.
- Total: Total of all reporting groups
Arm/Group | Bilateral Priming | Health Education | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change Score of Chedoke Arm and Hand Activity Index Nine (CAHAI 9) Baseline to Follow-up (2 Timepoints)
Description: The change score (Follow-up - Baseline) for the Chedoke Arm and Hand Activity Index 9 is reported. The change score scale ranges 0(min) to 63 (max). Higher scores indicate greater ability. Follow-up is at 6 weeks post treatment cessation. The scale measure bilateral activity performance.
Time Frame: value at 6 weeks minus value at baseline
Population: individuals who have survived a stroke greater than 6 months prior to enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bilateral Priming | Health Education
Number analyzed (Participants) | 7 | 7
score on a scale | 6.69 (1.2) | 5.03 (1.8)

2. Secondary Outcome: Change Score (Value at Follow-up - Value at Baseline) Fugl Meyer Upper Extremity Test of Function
Description: Change score between 2-time points (6 weeks follow up - baseline) Change score scale: minimum is 0 and maximum is 66. Higher scores indicate better outcomes.
Time Frame: value at 6 weeks minus value at baseline
Population: individuals who have survived a stroke greater than 6 months prior to enrollment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Bilateral Priming | Health Education
Number analyzed (Participants) | 7 | 7
units on a scale | 10 (2.5) | 4.3 (1.67)

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events reported to IRB
Groups:
- Bilateral Priming: Experimental group: There are 2 parts to this behavioral intervention. Bilateral priming and task specific training Dosage: 15 minutes of bilateral priming per day 3/days per week for 5/wks. Also 45 minutes of task specific training is delivered 3/days per week for 5/wks. The total of 30 hours can be completed within 6 weeks.
  Dosage frequency 2 times per day. Dosage type: Research participant must perform activities with affected hand (bilateral priming and task specific training) as directed by an occupational therapist
  rec
- Health Care Education: Active comparator : There are 2 parts to this behavioral intervention. Education on stroke health issues and task specific training. Health care education comes in the form of on-line games.
  Dosage: 15 minutes per day of computerized education 3/days per week for 5/wks. Also 45 minutes of task specific training is delivered 3/days per week for 5/wks. The total of 30 hours can be completed within 6 weeks.
  Dosage frequency 2 times per day for both parts of intervention Dosage type: Research participant must perform computerized education games as well as activities with the affected hand as directed by an occupational therapist
Arm/Group | Bilateral Priming | Health Care Education
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bilateral Priming (N=8) | Health Care Education (N=8)
Hospitalization (Infections and infestations) | 1 (1) | 0 (0) — A hospitalization was required that was not related to research protocol or the body system that the research was addressing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No